CLINICAL TRIAL: NCT00560755
Title: An Open-label, Multi-centre Study of the Safety of a 2-dose Regimen of a Combined Measles, Mumps, Rubella and Varicella Live Vaccine (ProQuad®) Manufactured With Recombinant Human Albumin (rHA) When Administered to Children in Their Second Year of Life
Brief Title: Safety Study of ProQuad® rHA in Infants (V221-037)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V221-037; MRV01C (Other: Sanofi Pasteur MSD Protocol Number); 2007-002438-12 (EudraCT Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Measles; Mumps; Rubella; Varicella
Keywords: Prevention of: measles, mumps, rubella and varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ProQuad® (Experimental): Healthy infants (12 to 22 months of age) received 2 doses of ProQuad® (Dose 1 on Day 1 and Dose 2 on Day 28 to 42) via subcutaneous injection into the deltoid muscle.
  Interventions: Biological: ProQuad®

INTERVENTIONS:
Biological: ProQuad® — ProQuad® manufactured with recombinant human albumin (rHA) is an investigational combined attenuated live virus vaccine for vaccination against measles, mumps, rubella and varicella viruses.

SUMMARY:
Primary objective: To describe the safety profile of a second dose of ProQuad® manufactured with recombinant human albumin (rHA) when administered to children in their second year of life.

Secondary objectives: To describe the safety profile of a first dose of ProQuad® manufactured with rHA when administered to children in their second year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject of either gender,
* Age from 12 to 22 months,
* Negative clinical history of infection with measles, mumps, rubella, varicella or zoster,
* Informed consent form signed by the parent(s) or by legal representative
* Parent(s) or legal representative able to attend all schedule visits with the subject and to understand and comply with the study procedures

Exclusion Criteria:

* Recent (≤ 3 days) history of febrile illness
* Prior receipt of measles, mumps, rubella and/or varicella vaccination, either alone or in any combination
* Recent (≤ 30 days) exposure to measles, mumps, rubella, varicella or zoster
* Prior known sensitivity/allergy to any component of the vaccine
* Severe chronic disease,
* Blood dyscrasias, leukaemia, lymphomas of any type, or other malignant neoplasms affecting the haematopoietic and lymphatic system
* Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection
* Humoral or cellular immunodeficiency,
* Current immunosuppressive therapy
* Family history of congenital or hereditary immunodeficiency
* Hereditary problems of fructose intolerance
* Known personal history of encephalopathy, seizure disorder or progressive, evolving or unstable neurological condition,
* Known active tuberculosis
* Recent (≤ 2 days) tuberculin test or scheduled tuberculin test through Visit 3
* Receipt of immunoglobulins or blood-derived products in the past 150 days
* Receipt of an inactivated vaccine in the past 14 days
* Receipt of a live vaccine in the past 28 days
* Any medical condition which, in the opinion of the investigator, might interfere with the evaluation of study objectives
* Participation in another clinical study in the past 30 days

Ages: 12 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3388 (Actual)
Dates: Start 2007-10-24 (Actual); Primary Completion 2008-11-24 (Actual); Study Completion 2008-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne FIQUET, MD, Study Director — MCM Vaccines B.V.

REFERENCES:
- [Derived] Ruger G, Gabutti G, Rumke H, Rombo L, Bernaola E, Diez-Domingo J, Martinon-Torres F, Hogh B, Konstantopoulos A, Fiquet A, Thomas S, Eymin C, Baudin M. Safety of a 2-dose regimen of a combined measles, mumps, rubella and varicella live vaccine manufactured with recombinant human albumin. Pediatr Infect Dis J. 2012 Nov;31(11):1166-72. doi: 10.1097/INF.0b013e318267fd8b. PMID 22772170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy pediatric participants were enrolled at 84 study centers in 7 European countries.
Period: Overall Study
Arm/Group | ProQuad®
Started | 3388 (Vaccinated (at least one ProQuad® dose))
ProQuad® Dose 1 and Dose 2 | 3346
Completed | 3328
Not Completed | 60
Not completed — Protocol Violation | 15
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 9
Not completed — Adverse Event | 8
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | ProQuad®
Number analyzed (Participants) | 3388
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1650
  Male | 1738

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) After ProQuad® Dose 2
Description: The percentage of participants experiencing an AE(s) for up to 28 days after the second ProQuad® injection was determined.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 57.66 [55.96 to 59.34]

2. Primary Outcome: Percentage of Participants Experiencing a Vaccine-related AE After ProQuad® Dose 2
Description: The percentage of participants experiencing a vaccine-related AEs for up to 28 days after the second ProQuad® injection was determined.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 41.77 [40.09 to 43.47]

3. Primary Outcome: Percentage of Participants Experiencing a Solicited Injection-site AE After ProQuad® Dose 2
Description: The solicited injection-site AEs erythema, swelling, and pain were monitored for 4 days after administration of ProQuad® Dose 2.
Time Frame: Up to Day 46 (for 4 days following ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants
  Injection-site erythema | 30.46 [28.90 to 32.05]
  Injection-site swelling | 13.23 [12.09 to 14.42]
  Injection-site pain | 11.49 [10.43 to 12.62]

4. Primary Outcome: Percentage of Participants Experiencing a Unsolicited Injection-site AE After ProQuad® Dose 2
Description: The percentage of participants experiencing a unsolicited injection-site AE(s) were monitored for up to 28 days after the second ProQuad® injection.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 1.65 [1.24 to 2.14]

5. Primary Outcome: Percentage of Participants Experiencing a Injection-site Rash of Interest AE After ProQuad® Dose 2
Description: Injection-site rashes of interest, including measles-like, rubella-like, and vesicular, were monitored for up to 28 days after the second ProQuad® injection.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 0.03 [0.00 to 0.17]

6. Primary Outcome: Percentage of Participants Experiencing a Systemic AE After ProQuad® Dose 2
Description: Systemic AEs were monitored for up to 28 days after the second ProQuad® injection.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 40.42 [38.76 to 42.11]

7. Primary Outcome: Percentage of Participants Experiencing a Vaccine-related Systemic AE After ProQuad® Dose 2
Description: Vaccine-related systemic AEs were monitored for up to 28 days after the second ProQuad® injection.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 13.44 [12.30 to 14.64]

8. Primary Outcome: Percentage of Participants Experiencing a Non-injection-site Rash of Interest AE After ProQuad® Dose 2
Description: Non-injection-site rashes of interest, including measles-like, rubella-like, varicella-like, and zoster-like rashes, were monitored for up to 28 days after the second ProQuad® injection.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants
  Measles-like rash | 1.62 [1.22 to 2.10]
  Rubella-like rash | 0.57 [0.34 to 0.89]
  Varicella-like rash | 0.63 [0.39 to 0.96]
  Zoster-like rash | 0.03 [0.00 to 0.17]

9. Primary Outcome: Percentage of Participants Experiencing a Mumps-like Illness After ProQuad® Dose 2
Description: The percentage of participants experiencing a mumps-like illness for up to 28 days after the second ProQuad® injection was determined.
Time Frame: Up to Day 70 (up to 28 days after ProQuad® Dose 2)
Population: All participants who received the second ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 0.03 [0.00 to 0.17]

10. Primary Outcome: Percentage of Participants Experiencing a Serious AE (SAE) After ProQuad® Dose 2
Description: Serious AEs ere defined as any untoward consequence that results in death, is life-threatening, requires hospitalization or prolongs existing hospitalization, is a congenital anomaly/birth defect, or is any other medically important event.
Time Frame: Up to Day 84 (up to 42 days after ProQuad® Dose 2)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 0.66 [0.41 to 0.99]

11. Primary Outcome: Percentage of Participants Experiencing a Vaccine-related SAE After ProQuad® Dose 2
Description: Vaccine-related SAEs were defined as any untoward consequence that results in death, is life-threatening, requires hospitalization or prolongs existing hospitalization, is a congenital anomaly/birth defect, or is any other medically important event.
Time Frame: Up to Day 84 (up to 42 days after ProQuad® Dose 2)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3342
Percentage of Participants | 0.21 [0.08 to 0.43]

12. Secondary Outcome: Percentage of Participants Experiencing a Solicited Injection-site AE After ProQuad® Dose 1
Description: The solicited injection-site AEs erythema, swelling, and pain were monitored for 4 days after administration of ProQuad® Dose 1.
Time Frame: From Day 1 to Day 4 (for 4 days following ProQuad® Dose 1)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3376
Percentage of Participants
  Injection-site erythema | 14.31 [13.14 to 15.53]
  Injection-site swelling | 5.57 [4.82 to 6.40]
  Injection-site pain | 10.31 [9.30 to 11.38]

13. Secondary Outcome: Percentage of Participants Experiencing a Unsolicited Injection-site AE After ProQuad® Dose 1
Description: Unsolicited injection-site AEs were monitored for up to 28 days after the first ProQuad® injection.
Time Frame: Up to Day 28 (28 days after ProQuad® Dose 1)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3376
Percentage of Participants | 7.43 [6.57 to 8.37]

14. Secondary Outcome: Percentage of Participants With ≥ 1 Rectal Temperature Reading ≥ 38.0° C After ProQuad® Dose 1
Description: The percentage of participants with at least 1 rectal temperature reading ≥ 38.0° C was determined.
Time Frame: Up to Day 28 (28 days after ProQuad® Dose 1)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3376
Percentage of Participants | 56.10 [0.85 to 1.61]

15. Secondary Outcome: Percentage of Participants Experiencing a Systemic AE After ProQuad® Dose 1
Description: Systemic AEs were monitored for up to 28 days after the first ProQuad® injection.
Time Frame: Up to Day 28 (28 days after ProQuad® Dose 1)
Population: All participants who received the first ProQuad® dose and had safety follow-up data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ProQuad®
Number analyzed (Participants) | 3376
Percentage of Participants | 64.10 [62.45 to 65.72]

ADVERSE EVENTS:
Time Frame: ProQuad® Dose 1: Up to Day 28 ProQuad® Dose 2: Up to Day 84 (up to 42 days after Dose 2)
Description: Participants who were vaccinated and have safety follow-up data are included. Data are presented separately for each post-dose monitoring period.
Groups:
- ProQuad® Arm: Dose 2: Healthy infants (12 to 22 months of age) received ProQuad® Dose 2 on Day 28 to Day 42.
- ProQuad® Arm: Dose 1: Healthy infants (12 to 22 months of age) received ProQuad® Dose 1 on Day 1.
Arm/Group | ProQuad® Arm: Dose 2 | ProQuad® Arm: Dose 1
Serious Adverse Events (participants affected / at risk) | 22/3342 | 40/3376
Other Adverse Events (participants affected / at risk) | 1507/3342 | 2057/3376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProQuad® Arm: Dose 2 (N=3342) | ProQuad® Arm: Dose 1 (N=3376)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 6 (6)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 6 (6) | 10 (10)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Norwalk virus (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pseudocroup (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsilitis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProQuad® Arm: Dose 2 (N=3342) | ProQuad® Arm: Dose 1 (N=3376)
Injection site erythema (General disorders) | 1024 (1032) | 628 (664)
Injection site pain (General disorders) | 384 (385) | 351 (352)
Injection site swelling (General disorders) | 447 (449) | 225 (228)
Pyrexia (General disorders) | 526 (591) | 1122 (1274)
Nasopharyngitis (Infections and infestations) | 174 (184) | 185 (198)
Diarrhoea (Gastrointestinal disorders) | 111 (120) | 191 (207)
Rhinits (Infections and infestations) | 142 (148) | 181 (198)
Cough (Respiratory, thoracic and mediastinal disorders) | 166 (178) | 199 (211)
Rash (Skin and subcutaneous tissue disorders) | 101 (103) | 226 (235)
Rash mobilliform (Skin and subcutaneous tissue disorders) | 54 (55) | 232 (236)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sanofi Pasteur MSD shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).